CLINICAL TRIAL: NCT02281825
Title: Correlating Real and Virtual World Behavioral Fluctuations in Adolescence
Status: Completed | Type: Observational
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Sponsor
Other Study IDs: sha-0001-14
Record Dates: First submitted 2014-10-29; First posted 2014-11-04 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Attention-Deficit and Hyperactivity Disorder; Anxiety; Disruptive Mood Dysregulation Disorder; Depression; Oppositional Defiant Disorder; Conduct
Keywords: Attention-Deficit and Hyperactivity Disorder; Anxiety; Impulsivity; Computer Games; Depression
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Anxiety Disorders; Depression; Oppositional Defiant Disorder; Behavior; Impulsive Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Adolescents without any psychiatric disorder
- Study: Adolescents with psychiatric disorder of the following: Attention-Deficit and Hyperactivity Disorder, Conduct, Oppositional defiant Disorder, Anxiety, Depression, Disruptive Mood Dysregulation Disorder

SUMMARY:
The present study will explore a new approach to ongoing evaluation and monitoring of fluctuations in personality traits via commercial video games. The aim of this longitudinal study is to examine the influence of everyday life event on video games performance as a function of individual differences in gaming behavioral patterns. focusing on the ongoing performance vacillations of the patient on commercial video games will offer insights in to possibly new generation of real time assessment medium of ongoing behavior.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will have normal or corrected to normal vision with no sensory/motor disturbance
* An accessible computer at the house hold
* Previous experience in playing computer games.

Exclusion Criteria:

* drug abuse
* head injury
* living in a boarding school and a major psychiatric or neurological disorder.

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Male adolescents, 13-18, with and without psychopathology, evaluated and diagnosed by psychiatrists. Adolescents will be recruited from Shalvata MHC children and adolescents outpatient clinic and from convinience sample in the community.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Impulsivity manifested within game-play | 3 weeks
  In-Game kill/Stealth ratio
Activity manifested within game-play | 3 weeks
  In-Game number of missions and sub-mission attained
Aggresion manifested within game-play | 3 weeks
  In-Game aimed killing

CONTACTS AND LOCATIONS:
Overall Officials: Aviv Segev, MD, Principal Investigator — Shalvata MHC, Sackler Faculty of Medicine, TA Uni.
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel